CLINICAL TRIAL: NCT04851938
Title: Evaluation of the Effect of Transcutaneous Electrical Nerve Stimulation Applied In Different Frequencies on Hormone Levels, Birth Pain Perception and Anxiety During Delivery
Brief Title: Evaluation of the Effect of Transcutaneous Electrical Nerve Stimulation During Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Rukiye Sülü, Health Sciences Faculty Midwifery Department, Cukurova University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CukurovaU TYL-2020-12916
Record Dates: First submitted 2021-04-10; First posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Anxiety, Hormone, Labour, Pain, Midwife, Pregnant, Transcutaneous Electrical Nerve Stimulation
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active TENS 1 Group (Active Comparator)
  Interventions: Device: transcutaneous electrical nerve stimulation device
- Active TENS 2 Group (Active Comparator)
  Interventions: Device: transcutaneous electrical nerve stimulation device
- Placebo Group (Placebo Comparator)
  Interventions: Device: transcutaneous electrical nerve stimulation device
- Control Group (Sham Comparator)
  Interventions: Device: transcutaneous electrical nerve stimulation device

INTERVENTIONS:
Device: transcutaneous electrical nerve stimulation device — The application of transcutaneous electrical nerve stimulation is a nonpharmacological method that midwives can apply and determining the effect on these factors will be a guide for the future applications.

SUMMARY:
Pain and anxiety levels experienced during labour are important factors affecting mother and baby health. An indicator that affects these factors is the levels of hormones that special for birth in the mother's blood. The application of transcutaneous electrical nerve stimulation is a nonpharmacological method that midwives can apply and determining the effect on these factors will be a guide for the future applications.

The research will be conducted between 20 March 2020 and 10 March 2021 at the Adana Seyhan State Hospital of the Ministry of Health of the Republic of Turkiye. The universe will be formed by the all pregnant women who are accepted to give birth to the birth room of the named hospital. The number of normal births in the relevant hospital in 2019 is 5979 per year. Power analysis was done with Gpower 3.1 for the number of samples. Báez-Suárez et al. Based on his study, the standard deviation of the pain scale was found as 1.48 and it was determined that at least 25 pregnant women per group with %5 error and %90 strength would be sufficient. It was planned to conduct a study with 28 pregnant women per group, with an increase in the sample size by %10, with the prospect of possible employment. One hundred and twelve pregnant women selected among pregnant women will be divided into 4 groups using a simple randomisation method and a random sequence will be created. Active transcuteneous electrical nerve stimulation at different doses will be applied to the two groups and the third group will be set as a placebo group. In the active phases of labour, active trancutaneous electrical nerve stimulation, which is adjusted to the first group of the pregnant women with a cervical aperture of at least 4 cm, modified biphasic asymmetric pulseand it was set to a pulse width of 100 μs and a frequency of 100 Hz (1). In the active transcutaneous electrical nerve stimulation second group, it emitted an asyymetric, balanced, biphasic square waveform at a mixed stimulating frequency that randomly varied between 80 and 100 Hz, and it had a pulse duration of 350 μs (2) will be applied for 30 minutes. Transcutaneous electrical nerve stimulation electrodes will be connected to the placebo group and 30 minutes will be waited without electric application. Transcutaneous electrical nerve stimulation electrodes will be connected to the control group and 30 minutes will be waited without electric application. Transcutaneous electrical nerve stimulation will be connected to the spinal cord in parallel with the levels of T10-L1 and S2-4 with two adhesive electrodes. Before and after transcutaneous electrical nerve stimulation application to pregnant women, hormon levels, visual analogue scale (VAS), pain assessment, state worry scale for anxiety assessment will be performed. Statistical Package for the Social Sciences 20.0 program will be used in the analysis of the data.

Birth pain is one of the most common types of pain. Various studies have been conducted on whether or not birth pain can be effectively reduced with transcutaneous electrical nerve stimulation application. However, no study evaluating the effect of transcutaneous electrical nerve stimulation application at different frequencies during delivery as a placebo controlled and double blind experimental study in terms of perception of birth pain, anxiety, hormon levels such as endrophin, oxytocin and cortisol was not found. Therefore, this study will be conducted as a randomised controlled experimental study to evaluate the effect of transcutaneous electrical nerve stimulation on birth pain, endorphine level, anxiety and satisfaction during delivery.

ELIGIBILITY:
Inclusion Criteria:

* 38-42 "week of pregnancy"
* Who will give normal vaginal delivery
* Dilatation of 4 cm and above
* Single fetus and head presentation
* Can speak Turkish and communicate
* Agreeing to participate in the study
* Not having risky pregnancy

Exclusion Criteria:

* Application of induction
* Using birth analgesia / anesthesia
* With pacemakers
* With skin damage in the area where TENS will be applied
* With any skin disease
* With contraction anomalies
* With epilepsy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2020-03-20 (Actual); Primary Completion 2021-05-20 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
pain perception and anxiety | 30 minutes
  Pain and anxiety levels experienced during labour are important factors affecting mother and baby health. For pain perseption VAS scale was used. For anxiety state anxiety scale was used.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Sarıcam, Turkey (Türkiye)